CLINICAL TRIAL: NCT03972813
Title: Optimizing HPV Vaccine Introduction in Shanghai, China
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19, we were unable to continue data collection in China.
Sponsor: University of Michigan (Other)
Collaborators: Shanghai Municipal Center for Disease Control and Prevention (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Abram Wagner, Research Assistant Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HUM00155864; K01AI137123 (NIH)
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Vaccine Refusal
Keywords: HPV Vaccines; China
MeSH Terms: conditions — Vaccination Refusal

STUDY DESIGN:
Intervention Model Description: In this educational intervention, there are three dimensions of variability: cancer messaging, communicability messaging, and age messaging. For cancer messaging there are two possibilities: one message focused more on cervical cancer, one message on cancer in general. For communicability, one message will have information on sexual transmission, a second on infectiousness in general, and a third will have no information about communicability. For age, one will mention that the vaccine is available for 9-45 year olds, the second will mention that and additionally recommend children 11 years old to receive the vaccine, and the third will recommend children 18 years old to receive the vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- cervical cancer - sexually transmitted (STD) - standard (Experimental): The Human Papilloma Virus (HPV) causes cervical cancer. HPV is a sexually transmitted disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China.
  Interventions: Behavioral: Information about STDs; Behavioral: Standard age information; Behavioral: Cervical cancer
- cervical cancer - STD - 12 years old (y.o.) (Experimental): The Human Papilloma Virus (HPV) causes cervical cancer. HPV is a sexually transmitted disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between grade school and middle school is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Information about STDs; Behavioral: Recommendation for children 12 years old; Behavioral: Cervical cancer
- cervical cancer - STD - 18 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cervical cancer. HPV is a sexually transmitted disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between high school and college or work is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Information about STDs; Behavioral: Recommendation for children 18 years old; Behavioral: Cervical cancer
- cervical cancer - infectious - standard (Experimental): The Human Papilloma Virus (HPV) causes cervical cancer. HPV is an infectious disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China.
  Interventions: Behavioral: Information about infectious disease; Behavioral: Standard age information; Behavioral: Cervical cancer
- cervical cancer - infectious - 12 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cervical cancer. HPV is an infectious disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between grade school and middle school is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Information about infectious disease; Behavioral: Recommendation for children 12 years old; Behavioral: Cervical cancer
- cervical cancer - infectious - 18 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cervical cancer. HPV is an infectious disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between high school and college or work is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Information about infectious disease; Behavioral: Recommendation for children 18 years old; Behavioral: Cervical cancer
- cervical cancer - blank - standard (Experimental): The Human Papilloma Virus (HPV) causes cervical cancer. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China.
  Interventions: Behavioral: Standard age information; Behavioral: Cervical cancer; Behavioral: Blank information about communicability
- cervical cancer - blank - 12 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cervical cancer. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between grade school and middle school is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Recommendation for children 12 years old; Behavioral: Cervical cancer; Behavioral: Blank information about communicability
- cervical cancer - blank - 18 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cervical cancer. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between high school and college or work is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Recommendation for children 18 years old; Behavioral: Cervical cancer; Behavioral: Blank information about communicability
- many cancers - STD - standard (Experimental): The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is a sexually transmitted disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China.
  Interventions: Behavioral: Broadened information about cancers; Behavioral: Information about STDs; Behavioral: Standard age information
- many cancers - STD - 12 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is a sexually transmitted disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between grade school and middle school is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Broadened information about cancers; Behavioral: Information about STDs; Behavioral: Recommendation for children 12 years old
- many cancers - STD - 18 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is a sexually transmitted disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between high school and college or work is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Broadened information about cancers; Behavioral: Information about STDs; Behavioral: Recommendation for children 18 years old
- many cancers - infectious - standard (Experimental): The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is an infectious disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China.
  Interventions: Behavioral: Broadened information about cancers; Behavioral: Information about infectious disease; Behavioral: Standard age information
- many cancers - infectious - 12 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is an infectious disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between grade school and middle school is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Broadened information about cancers; Behavioral: Information about infectious disease; Behavioral: Recommendation for children 12 years old
- many cancers - infectious - 18 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is an infectious disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between high school and college or work is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Broadened information about cancers; Behavioral: Information about infectious disease; Behavioral: Recommendation for children 18 years old
- many cancers - blank - standard (Experimental): The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China.
  Interventions: Behavioral: Broadened information about cancers; Behavioral: Standard age information; Behavioral: Blank information about communicability
- many cancers - blank - 12 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between grade school and middle school is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Broadened information about cancers; Behavioral: Recommendation for children 12 years old; Behavioral: Blank information about communicability
- many cancers - blank - 18 y.o. (Experimental): The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between high school and college or work is a particularly good time to think about the HPV vaccine.
  Interventions: Behavioral: Broadened information about cancers; Behavioral: Recommendation for children 18 years old; Behavioral: Blank information about communicability

INTERVENTIONS:
Behavioral: Broadened information about cancers — Caregivers receive information that HPV causes more than just cervical cancer.
  Arms: many cancers - STD - 12 y.o.; many cancers - STD - 18 y.o.; many cancers - STD - standard; many cancers - blank - 12 y.o.; many cancers - blank - 18 y.o.; many cancers - blank - standard; many cancers - infectious - 12 y.o.; many cancers - infectious - 18 y.o.; many cancers - infectious - standard
Behavioral: Information about STDs — Caregivers learn that HPV is an STD.
  Arms: cervical cancer - STD - 12 years old (y.o.); cervical cancer - STD - 18 y.o.; cervical cancer - sexually transmitted (STD) - standard; many cancers - STD - 12 y.o.; many cancers - STD - 18 y.o.; many cancers - STD - standard
Behavioral: Information about infectious disease — Caregivers learn that HPV is infectious (but information that it is an STD is omitted).
  Arms: cervical cancer - infectious - 12 y.o.; cervical cancer - infectious - 18 y.o.; cervical cancer - infectious - standard; many cancers - infectious - 12 y.o.; many cancers - infectious - 18 y.o.; many cancers - infectious - standard
Behavioral: Recommendation for children 12 years old — Caregivers are prompted to get their child vaccinated when the child is 12 years old.
  Arms: cervical cancer - STD - 12 years old (y.o.); cervical cancer - blank - 12 y.o.; cervical cancer - infectious - 12 y.o.; many cancers - STD - 12 y.o.; many cancers - blank - 12 y.o.; many cancers - infectious - 12 y.o.
Behavioral: Recommendation for children 18 years old — Caregivers are prompted to get their child vaccinated when the child is 18 years old.
  Arms: cervical cancer - STD - 18 y.o.; cervical cancer - blank - 18 y.o.; cervical cancer - infectious - 18 y.o.; many cancers - STD - 18 y.o.; many cancers - blank - 18 y.o.; many cancers - infectious - 18 y.o.
Behavioral: Standard age information — Caregivers are given information about when the HPV vaccination can be given in China, but no additional recommendations.
  Arms: cervical cancer - blank - standard; cervical cancer - infectious - standard; cervical cancer - sexually transmitted (STD) - standard; many cancers - STD - standard; many cancers - blank - standard; many cancers - infectious - standard
Behavioral: Cervical cancer — Caregivers are told that HPV causes cervical cancer.
  Arms: cervical cancer - STD - 12 years old (y.o.); cervical cancer - STD - 18 y.o.; cervical cancer - blank - 12 y.o.; cervical cancer - blank - 18 y.o.; cervical cancer - blank - standard; cervical cancer - infectious - 12 y.o.; cervical cancer - infectious - 18 y.o.; cervical cancer - infectious - standard; cervical cancer - sexually transmitted (STD) - standard
Behavioral: Blank information about communicability — Caregivers are not given any information on how HPV is spread.
  Arms: cervical cancer - blank - 12 y.o.; cervical cancer - blank - 18 y.o.; cervical cancer - blank - standard; many cancers - blank - 12 y.o.; many cancers - blank - 18 y.o.; many cancers - blank - standard

SUMMARY:
Within low, middle, and upper income countries, low vaccine coverage results from both obstacles to vaccine access and low confidence in vaccine programs. Thus, it is critical to determine how best to enhance trust in vaccines as increasing numbers of vaccines are recommended for use. Even though the context accompanying the initial roll-out of a vaccine can have a large impact on people's perceptions of the vaccine and the corresponding disease, it is not clear how to best introduce a vaccine to increase public confidence and enhance uptake. The US roll-out of the human papillomavirus (HPV) vaccine framed HPV as a sexually transmitted infection, which proved to be an impediment to efforts to increase vaccine uptake >10 years after its introduction. This study will use an educational experiment, where parents of children will be exposed to information about the HPV vaccination in different ways. Parents will be introduced to the HPV vaccine through different scenarios with varying emphases (i.e., age at vaccination, types of transmission, type of cancer prevention). The aim will be to determine how the framing of the HPV vaccination across several dimensions affects short-term willingness to receive it.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children 2-18 years old.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1021 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abram L Wagner, PhD, MPH, Principal Investigator — University of Michigan
Locations (1):
- Shanghai CDC, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be uploaded to a public repository after each wave of data collection is complete.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Wave 1 (aim 1): data available end of 2019
Access Criteria: The data is freely and publicly available
URL: https://doi.org/10.6084/m9.figshare.12980042

REFERENCES:
- [Result] Huang Z, Ji M, Ren J, Sun X, Boulton ML, Zikmund-Fisher BJ, Wagner AL. Effect of the framing of HPV vaccination on parents' willingness to accept an HPV vaccine. Vaccine. 2022 Feb 7;40(6):897-903. doi: 10.1016/j.vaccine.2021.12.051. Epub 2022 Jan 4. PMID 34996644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: summer 2019 Recruitment locations: immunization clinics and schools in 40 townships in Shanghai, China
Groups:
- Many Cancers - STD - Standard: The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is a sexually transmitted disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China.
  Broadened information about cancers: Caregivers receive information that HPV causes more than just cervical cancer.
  Information about STDs: Caregivers learn that HPV is an STD.
  Standard age information: Caregivers are given information about when the HPV vaccination can be given in China, but no additional recommendations.
- Many Cancers - STD - 12 y.o.: The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is a sexually transmitted disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between grade school and middle school is a particularly good time to think about the HPV vaccine.
  Broadened information about cancers: Caregivers receive information that HPV causes more than just cervical cancer.
  Information about STDs: Caregivers learn that HPV is an STD.
  Recommendation for children 12 years old: Caregivers are prompted to get their child vaccinated when the child is 12 years old.
- Many Cancers - STD - 18 y.o.: The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is a sexually transmitted disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between high school and college or work is a particularly good time to think about the HPV vaccine.
  Broadened information about cancers: Caregivers receive information that HPV causes more than just cervical cancer.
  Information about STDs: Caregivers learn that HPV is an STD.
  Recommendation for children 18 years old: Caregivers are prompted to get their child vaccinated when the child is 18 years old.
- Many Cancers - Infectious - Standard: The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is an infectious disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China.
  Broadened information about cancers: Caregivers receive information that HPV causes more than just cervical cancer.
  Information about infectious disease: Caregivers learn that HPV is infectious (but information that it is an STD is omitted).
  Standard age information: Caregivers are given information about when the HPV vaccination can be given in China, but no additional recommendations.
- Many Cancers - Infectious - 12 y.o.: The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is an infectious disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between grade school and middle school is a particularly good time to think about the HPV vaccine.
  Broadened information about cancers: Caregivers receive information that HPV causes more than just cervical cancer.
  Information about infectious disease: Caregivers learn that HPV is infectious (but information that it is an STD is omitted).
  Recommendation for children 12 years old: Caregivers are prompted to get their child vaccinated when the child is 12 years old.
- Many Cancers - Infectious - 18 y.o.: The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  HPV is an infectious disease. Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between high school and college or work is a particularly good time to think about the HPV vaccine.
  Broadened information about cancers: Caregivers receive information that HPV causes more than just cervical cancer.
  Information about infectious disease: Caregivers learn that HPV is infectious (but information that it is an STD is omitted).
  Recommendation for children 18 years old: Caregivers are prompted to get their child vaccinated when the child is 18 years old.
- Many Cancers - Blank - Standard: The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China.
  Broadened information about cancers: Caregivers receive information that HPV causes more than just cervical cancer.
  Standard age information: Caregivers are given information about when the HPV vaccination can be given in China, but no additional recommendations.
  Blank information about communicability: Caregivers are not given any information on how HPV is spread.
- Many Cancers - Blank - 12 y.o.: The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between grade school and middle school is a particularly good time to think about the HPV vaccine.
  Broadened information about cancers: Caregivers receive information that HPV causes more than just cervical cancer.
  Recommendation for children 12 years old: Caregivers are prompted to get their child vaccinated when the child is 12 years old.
  Blank information about communicability: Caregivers are not given any information on how HPV is spread.
- Many Cancers - Blank - 18 y.o.: The Human Papilloma Virus (HPV) causes cancers all over the body, from the head to the reproductive system.
  Currently, safe and effective HPV vaccines are available for women 9-45 years of age in China. The transition between high school and college or work is a particularly good time to think about the HPV vaccine.
  Broadened information about cancers: Caregivers receive information that HPV causes more than just cervical cancer.
  Recommendation for children 18 years old: Caregivers are prompted to get their child vaccinated when the child is 18 years old.
  Blank information about communicability: Caregivers are not given any information on how HPV is spread.
Period: Overall Study
Arm/Group | Cervical Cancer - Sexually Transmitted (STD) - Standard | Cervical Cancer - STD - 12 Years Old (y.o.) | Cervical Cancer - STD - 18 y.o. | Cervical Cancer - Infectious - Standard | Cervical Cancer - Infectious - 12 y.o. | Cervical Cancer - Infectious - 18 y.o. | Cervical Cancer - Blank - Standard | Cervical Cancer - Blank - 12 y.o. | Cervical Cancer - Blank - 18 y.o. | Many Cancers - STD - Standard | Many Cancers - STD - 12 y.o. | Many Cancers - STD - 18 y.o. | Many Cancers - Infectious - Standard | Many Cancers - Infectious - 12 y.o. | Many Cancers - Infectious - 18 y.o. | Many Cancers - Blank - Standard | Many Cancers - Blank - 12 y.o. | Many Cancers - Blank - 18 y.o.
Started | 85 | 49 | 58 | 55 | 52 | 51 | 53 | 55 | 58 | 60 | 62 | 55 | 58 | 55 | 58 | 56 | 51 | 50
Completed (68 individuals completed the survey but did not answer the outcome) | 79 | 45 | 52 | 51 | 48 | 49 | 49 | 52 | 53 | 58 | 57 | 51 | 55 | 52 | 56 | 50 | 48 | 48
Not Completed | 6 | 4 | 6 | 4 | 4 | 2 | 4 | 3 | 5 | 2 | 5 | 4 | 3 | 3 | 2 | 6 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Cancer - Sexually Transmitted (STD) - Standard | Cervical Cancer - STD - 12 Years Old (y.o.) | Cervical Cancer - STD - 18 y.o. | Cervical Cancer - Infectious - Standard | Cervical Cancer - Infectious - 12 y.o. | Cervical Cancer - Infectious - 18 y.o. | Cervical Cancer - Blank - Standard | Cervical Cancer - Blank - 12 y.o. | Cervical Cancer - Blank - 18 y.o. | Many Cancers - STD - Standard | Many Cancers - STD - 12 y.o. | Many Cancers - STD - 18 y.o. | Many Cancers - Infectious - Standard | Many Cancers - Infectious - 12 y.o. | Many Cancers - Infectious - 18 y.o. | Many Cancers - Blank - Standard | Many Cancers - Blank - 12 y.o. | Many Cancers - Blank - 18 y.o. | Total
Number analyzed (Participants) | 79 | 45 | 52 | 51 | 48 | 49 | 49 | 52 | 53 | 58 | 57 | 51 | 55 | 52 | 56 | 50 | 48 | 48 | 953
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [36 to 42] | 38 [32 to 41] | 39 [33.5 to 40.5] | 38 [32 to 42] | 35 [32 to 39] | 37.5 [35 to 43] | 39 [35 to 41] | 36 [32 to 40] | 37 [32 to 40] | 36 [33 to 40] | 37 [34 to 40] | 37 [32 to 41] | 37 [32 to 40] | 37 [35 to 40] | 37 [34 to 41] | 37 [35 to 40] | 38 [34 to 42] | 38 [34 to 41] | 37 [34 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 34 | 38 | 40 | 37 | 37 | 40 | 45 | 46 | 47 | 44 | 41 | 43 | 39 | 52 | 34 | 40 | 40 | 758
  Male | 18 | 11 | 14 | 11 | 11 | 12 | 9 | 7 | 7 | 11 | 13 | 10 | 12 | 13 | 4 | 16 | 8 | 8 | 195
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 79 | 45 | 52 | 51 | 48 | 49 | 49 | 52 | 53 | 58 | 57 | 51 | 55 | 52 | 56 | 50 | 48 | 48 | 953
Vaccinated at baseline [Count of Participants; unit: Participants] — Response to the question: "Has one of your children already received the HPV vaccine?"
  Participants | 4 | 4 | 2 | 1 | 4 | 6 | 2 | 3 | 2 | 3 | 4 | 2 | 3 | 3 | 3 | 2 | 2 | 3 | 53

OUTCOME MEASURES:

1. Primary Outcome: To Determine How the Framing of the HPV Vaccination Across Several Dimensions Affects Short-term Willingness to Receive it
Description: Immediately after the experimental component, parents will respond to the question "If you had a daughter, how willing would you be to give your daughter an HPV vaccine at 12 years of age?" This will be assessed on a 5-point scale from "not at all willing" (1) to "very willing" (5). The proportion of parents who select "somewhat" (4) or "very willing" (5) will be tallied as the primary outcome measure.
Time Frame: same day as intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Cervical Cancer - Sexually Transmitted (STD) - Standard | Cervical Cancer - STD - 12 Years Old (y.o.) | Cervical Cancer - STD - 18 y.o. | Cervical Cancer - Infectious - Standard | Cervical Cancer - Infectious - 12 y.o. | Cervical Cancer - Infectious - 18 y.o. | Cervical Cancer - Blank - Standard | Cervical Cancer - Blank - 12 y.o. | Cervical Cancer - Blank - 18 y.o. | Many Cancers - STD - Standard | Many Cancers - STD - 12 y.o. | Many Cancers - STD - 18 y.o. | Many Cancers - Infectious - Standard | Many Cancers - Infectious - 12 y.o. | Many Cancers - Infectious - 18 y.o. | Many Cancers - Blank - Standard | Many Cancers - Blank - 12 y.o. | Many Cancers - Blank - 18 y.o.
Number analyzed (Participants) | 79 | 45 | 52 | 51 | 48 | 49 | 49 | 52 | 53 | 58 | 57 | 51 | 55 | 52 | 56 | 50 | 48 | 48
Participants | 46 | 31 | 29 | 21 | 28 | 26 | 28 | 23 | 31 | 35 | 33 | 27 | 33 | 31 | 29 | 22 | 28 | 25

2. Secondary Outcome: To Determine How the Framing of the HPV Vaccination Across Several Dimensions Affects Sustained Willingness to Receive it
Description: Three years after the experimental component, parents will respond to the question "If you had a daughter, how willing would you be to give your daughter an HPV vaccine at 12 years of age?" This will be assessed on a 5-point scale from "not at all willing" (1) to "very willing" (5). The proportion of parents who select "somewhat" (4) or "very willing" (5) will be tallied as the primary outcome measure.
Time Frame: 3 years
Population: This study was terminated early because of COVID-19, and data on the secondary outcome were not collected.
Arm/Group | Cervical Cancer - Sexually Transmitted (STD) - Standard | Cervical Cancer - STD - 12 Years Old (y.o.) | Cervical Cancer - STD - 18 y.o. | Cervical Cancer - Infectious - Standard | Cervical Cancer - Infectious - 12 y.o. | Cervical Cancer - Infectious - 18 y.o. | Cervical Cancer - Blank - Standard | Cervical Cancer - Blank - 12 y.o. | Cervical Cancer - Blank - 18 y.o. | Many Cancers - STD - Standard | Many Cancers - STD - 12 y.o. | Many Cancers - STD - 18 y.o. | Many Cancers - Infectious - Standard | Many Cancers - Infectious - 12 y.o. | Many Cancers - Infectious - 18 y.o. | Many Cancers - Blank - Standard | Many Cancers - Blank - 12 y.o. | Many Cancers - Blank - 18 y.o.
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: This study is an educational/behavioral intervention. Any "physical" adverse event is not expected to occur. This study could change someone's attitude about the HPV vaccine for the worse - a behavioral/attitudinal adverse event.
  If acceptability of the vaccine is less than 40% (about 10% to 20% less than acceptability of what was found in previous studies), data collection will be temporarily stopped.
Arm/Group | Cervical Cancer - Sexually Transmitted (STD) - Standard | Cervical Cancer - STD - 12 Years Old (y.o.) | Cervical Cancer - STD - 18 y.o. | Cervical Cancer - Infectious - Standard | Cervical Cancer - Infectious - 12 y.o. | Cervical Cancer - Infectious - 18 y.o. | Cervical Cancer - Blank - Standard | Cervical Cancer - Blank - 12 y.o. | Cervical Cancer - Blank - 18 y.o. | Many Cancers - STD - Standard | Many Cancers - STD - 12 y.o. | Many Cancers - STD - 18 y.o. | Many Cancers - Infectious - Standard | Many Cancers - Infectious - 12 y.o. | Many Cancers - Infectious - 18 y.o. | Many Cancers - Blank - Standard | Many Cancers - Blank - 12 y.o. | Many Cancers - Blank - 18 y.o.
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/45 | 0/52 | 0/51 | 0/48 | 0/49 | 0/49 | 0/52 | 0/53 | 0/58 | 0/57 | 0/51 | 0/55 | 0/52 | 0/56 | 0/50 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/45 | 0/52 | 0/51 | 0/48 | 0/49 | 0/49 | 0/52 | 0/53 | 0/58 | 0/57 | 0/51 | 0/55 | 0/52 | 0/56 | 0/50 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/79 | 0/45 | 0/52 | 0/51 | 0/48 | 0/49 | 0/49 | 0/52 | 0/53 | 0/58 | 0/57 | 0/51 | 0/55 | 0/52 | 0/56 | 0/50 | 0/48 | 0/48

LIMITATIONS AND CAVEATS:
Note: Due to the COVID-19 pandemic, collection of data on the secondary outcome was stopped. Accordingly, the grant associated with this clinical trial had a change in scope.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT03972813/Prot_SAP_000.pdf